CLINICAL TRIAL: NCT04611022
Title: Intervention to Educate and Improve Underserved Populations' Uptake and Completion of the HPV Vaccine Series
Brief Title: Educate and Improve Underserved Populations' Uptake and Completion of the HPV Vaccine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-2236.cc; P30CA046934 (NIH)
Record Dates: First submitted 2020-09-30; First posted 2020-11-02 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Human Papilloma Virus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients Eligible for HPV Vaccine (Experimental)
  Interventions: Behavioral: HPV Educational Intervention

INTERVENTIONS:
Behavioral: HPV Educational Intervention — The videos are 8-minute narrative films created using an entertainment-education (E-E) approach that embeds an educational narrative message into an entertainment format such as media. E-E narratives have demonstrated a significant effect (r = .12, p < .001) on health behavior change. Evidence-based small media interventions that Dr. Borrayo has produced include videos that are highly verbal, visual, and entertaining (e.g., acted fictional stories). The aims of the video will be to model uptake of the HPV vaccine, but also to reinforce self-efficacy, subjective norms, and behavioral intentions, all significant precursors to behavior change.

SUMMARY:
The educational intervention to be delivered by the PN(Patient Navigator) consists of "toolkit education materials" developed by the National Cancer Institute (NCI) and a small media intervention (i.e., video) that our research team has developed. The NCI-produced toolkit education materials consist of Power Point presentations, flyers, and posters that contain information about HPV(Human Papilloma Virus), HPV-related cancers, and the importance of the HPV vaccine series for adolescents (9-17 years old) and young adults (18-26 year old) who are eligible for the vaccine.

DETAILED DESCRIPTION:
The investigator will use a one-group post-test design to assess the effects of the intervention on the primary outcomes. The educational intervention will be delivered to 400 participants by a trained CHE who will deliver the educational materials to eligible DHHA patients. The CHE will administer the post-education survey at baseline to participants. Additionally, we will use a one-group post-test design to assess the impact of the intervention on the secondary outcomes. At the patient-level, we will track participants that receive (a) 1st dose, 2nd dose, or 3rd dose of the HPV vaccine; and the number of referrals to care by recording the number of patients received (b) referrals to health insurance, discount, or no-cost HPV vaccine programs; or (c) to other services to facilitate HPV vaccine dose completion. To assess clinic-level impact, we will track each clinic's HPV vaccine rates for adolescents (9-17 years old) and young adults (18-26) and compare rates from before we start the intervention and then quarterly there after we have introduced the intervention to each respective Denver Health clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Be a Denver Health patient* 18-26 years old, who has not started or completed the HPV vaccine series (Vaccine completion for this age group is 3 doses).
2. Be a parent of a Denver Health adolescent patient* aged 9-17 years old, who has not started or completed the HPV vaccine series. (Vaccine completion is 2 doses for 9-14-year-old, and 3 doses for 14-17-year old)
3. English and/or Spanish Speaking
4. Stated willingness to comply with all study procedures and be available for the duration of the study

   * Denver Health patients will be identified from one of the following clinics; Denver Health Clinics Eastside Adult Clinic, Eastside Women's Care Clinic, Westside Adult Clinic, Westside Women's Care Clinic, Pavilion C: Women's Care Clinic, La Casa-Quigg Newton Family Health Center, Lowry Family Health Center, Montbello Family Health Center, Westwood Family Health Center, Parkhill Family Health Center, Webb Center For Primary Care, Pena Southwest Clinic

Exclusion Criteria:

1. Individuals who do not meet eligibility criteria, including individuals who do not speak English or Spanish [at the discretion of the CHE or PN upon recruitment]
2. Decisionally-challenged adults with cognitive or personality impairment or due to intoxication (alcohol or drugs) that might interfere with their ability to consent or participate in the study [at the discretion of the CHE or PN upon recruitment]
3. Individuals from vulnerable populations (e.g., inmates, homeless, pregnant women, and those with auditory impairment [at the discretion of the CHE or PN upon recruitment]
4. Individuals under the age of 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
The change in parents & young adults' knowledge & intentions to obtain the HPV vaccine | Day 0/Baseline
  Behavioral factors precede uptake of preventive vaccines. Measured by survey post watching HPV video.
Sociodemographic data (e.g., age, gender, ethnicity, insurance, income, zip code) as it relates to vaccine uptake | Day 0/Baseline
  Collected by the study team. Variables known as associated with vaccine uptake

SECONDARY OUTCOMES:
Uptake of one, two, or three HPV vaccine doses among adolescents (9 to 17 years old) and young adults (18-26 years old). | 3 and 6 months post intervention
  As determined by follow up phone calls. Number of vaccine doses are used to assess full protection (3 doses) or partial (<3 doses)

OTHER OUTCOMES:
Intervention's delivery and patient-level & system-level impact. | 3, 6, 9 and 12 months post intervention
  Interventions that can be delivered to impact patients & clinics are easier to implement. As determined by rates of HPV vaccine dose completion reported by clinics

CONTACTS AND LOCATIONS:
Overall Officials: Evelinn Borrayo, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT04611022/Prot_000.pdf
  • Informed Consent Form (2025-02-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT04611022/ICF_001.pdf